CLINICAL TRIAL: NCT02013167
Title: A Phase 3, Randomized, Open Label Study Investigating the Efficacy of the BiTE Antibody Blinatumomab Versus Standard of Care Chemotherapy in Adult Subjects With Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia (ALL) (TOWER Study)
Brief Title: Blinatumomab Versus Standard of Care Chemotherapy in Patients With Relapsed or Refractory Acute Lymphoblastic Leukemia (ALL)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00103311; 2013-000536-10 (EudraCT Number)
Record Dates: First submitted 2013-12-03; First posted 2013-12-17 (Estimated); Results first posted 2017-08-09 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Relapsed/Refractory B-precursor Acute Lymphoblastic Leukemia
Keywords: Relapsed; Refractory; B-precursor; Acute Lymphoblastic Leukemia; Philadelphia Negative; ALL; Blinatumomab; Leukemia; Standard of Care; SOC
MeSH Terms: conditions — Recurrence; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia | interventions — blinatumomab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Blinatumomab (Experimental): Participants received blinatumomab by continuous intravenous infusion (CIVI) over 4 weeks followed by a 2 week treatment-free interval for 2 induction cycles. Participants who achieved a bone marrow response, complete remission, or complete remission with partial or incomplete hematologic recovery (CR/CRh*/CRi) within 2 induction cycles of treatment could receive up to 3 additional consolidation cycles of blinatumomab.
  Participants who received 2 induction and up to 3 consolidation cycles of therapy and continued to have a bone marrow response or CR/CRh*/CRi could continue to receive blinatumomab for an additional 12 months (4 cycles), where 1 cycle consisted of 4 weeks of CIVI followed by an 8-week treatment-free period.
  The initial dose of blinatumomab was 9 μg/day for the first 7 days of treatment, increased to 28 μg/day starting on day 8 through day 29 and for all subsequent cycles.
  Interventions: Drug: Blinatumomab
- Standard of Care Chemotherapy (Active Comparator): Participants received one of four prespecified, investigator-chosen chemotherapy regimens for 2 induction cycles. Participants who achieved a bone marrow response, CR/CRh*/CRi within 2 induction cycles of treatment could receive up to 3 additional consolidation cycles of SOC chemotherapy.
  Participants who received 2 induction and up to 3 consolidation cycles of therapy and continued to have a bone marrow response or CR/CRh*/CRi could continue to receive SOC therapy for an additional 12 months.
  Interventions: Drug: Standard of Care Chemotherapy

INTERVENTIONS:
Drug: Blinatumomab — Blinatumomab is administered as a continuous intravenous infusion (CIV).
  Other Names: Blincyto®; AMG 103; MT103
  Arms: Blinatumomab
Drug: Standard of Care Chemotherapy — * FLAG (fludarabine, cytarabine arabinoside, and granulocyte colony-stimulating factor) ± anthracycline-based regimen (e.g. idarubicin 10 mg/m² days 1 & 3; fludarabine 30 mg/m² days 1-5; cytarabine arabinoside 2 g/m² days 1-5). Patients > 60 years: Idarubicin 5 mg/m² day 1 & 3; fludarabine 20 mg/m² day 1-5; cytarabine arabinoside 1 g/m² day 1-5
  * HiDAC (high-dose cytarabine arabinoside) - based regimen ≥1 g/m²/day ± anthracycline and/or in combination with other drugs such as native Escherichia coli asparaginase, polyethylene glycol linked to asparaginase (PEG-asparaginase), vinca alkaloids, steroids, etoposide or alkylating agents
  * High-dose methotrexate-based regimen (HDMTX; 500 mg/m² to 3 g/m² infused up to 24 hours) in combination with native E. coli asparaginase, PEG-asparaginase, vinca alkaloids, steroids, etoposide or alkylating agents.
  * Clofarabine as a single agent as recommended in the prescribing information or clofarabine-based regimens with 20 mg/m²/day for up to 5 days.
  Arms: Standard of Care Chemotherapy

SUMMARY:
The primary objective was to evaluate the effect of blinatumomab on overall survival when compared to standard of care (SOC) chemotherapy.

DETAILED DESCRIPTION:
Adults with relapsed/refractory B-cell precursor ALL were randomized in a 2:1 ratio to receive blinatumomab or 1 of 4 pre-specified, investigator-chosen, SOC chemotherapy regimens. Randomization was stratified by age (< 35 years vs ≥ 35 years of age), prior salvage therapy (yes vs no), and prior allogeneic HSCT (yes vs no) as assessed at the time of consent.

The study consisted of up to a 3-week screening and pre-phase period, a treatment period consisting of induction with 2 cycles of either blinatumomab or SOC chemotherapy, a consolidation phase of up to 3 additional cycles of protocol-specified therapy, and a maintenance phase for up to an additional 12 months with protocol-specified therapy. A safety follow-up visit 30 days after the last dose of protocol-specified therapy and a long-term follow-up period were included. The long-term follow-up part of the study was discontinued prematurely based on a recommendation from the data monitoring committee (DMC) that the study be stopped for benefit.

ELIGIBILITY:
* Subjects with Philadelphia negative B-precursor ALL, with any of the following:

  * refractory to primary induction therapy or refractory to salvage therapy,
  * in untreated first relapse with first remission duration <12 months
  * in untreated second or greater relapse
  * relapse at any time after allogeneic HSCT
* Subject has received intensive combination chemotherapy for the treatment of ALL for initial treatment or subsequent salvage therapy.
* Greater than 5% blasts in the bone marrow
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria

* Malignancy other than ALL within 5 years before blinatumomab treatment, except for adequately treated selected cancers without evidence of disease
* Diagnosis of Burkitt's leukemia according to World Health Organization classification, or human immunodeficiency virus (HIV), Hepatitis B or C, or other clinically significant disorder
* Current relevant central nervous system (CNS) pathology or known or suspected CNS involvement
* Isolated extramedullary disease
* Current autoimmune disease or history of autoimmune disease with potential CNS involvement
* Autologous HSCT within 6 weeks or allogeneic HSCT within 12 weeks before blinatumomab treatment, or eligibility for allogeneic HSCT at the time of enrollment
* Active acute grade 2 to 4 graft versus host disease (GvHD) according to Glucksberg et al (1974) criteria that required systemic treatment to prevent or treat GvHD 2 weeks before blinatumomab treatment
* Known exclusion criteria to investigator choice of SOC chemotherapy (per package insert)
* Cancer chemotherapy or radiotherapy with 2 weeks, or immunotherapy (included CD19 therapy) within 4 weeks of protocol-specified therapy
* Abnormal laboratory values (alanine or aspartate transaminase [ALT or AST] or alkaline phosphatase [ALP] ≥ 5 × upper limit of normal [ULN]; total bilirubin or creatinine ≥ 1.5 × ULN), or calculated creatinine clearance < 60 mL/min.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2014-01-03 (Actual); Primary Completion 2015-12-29 (Actual); Study Completion 2017-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (108):
- United States (15):
  - Research Site, Duarte, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Atlanta, Georgia
  - Research Site, Chicago, Illinois
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Rochester, Minnesota
  - Research Site, St Louis, Missouri
  - Research Site, New York, New York
  - Research Site, Durham, North Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Nashville, Tennessee
  - Research Site, Houston, Texas
  - Research Site, Milwaukee, Wisconsin
- Australia (6):
  - Research Site, St Leonards, New South Wales
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Parkville, Victoria
  - Research Site, Prahran, Victoria
  - Research Site, Murdoch, Western Australia
- Austria (3):
  - Research Site, Salzburg
  - Research Site, Vienna
  - Research Site, Wels
- Belgium (6):
  - Research Site, Antwerp
  - Research Site, Bruges
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Leuven
  - Research Site, Yvoir
- Bulgaria (2):
  - Research Site, Plovdiv
  - Research Site, Sofia
- Canada (2):
  - Research Site, Toronto, Ontario
  - Research Site, Montreal, Quebec
- Czechia (3):
  - Research Site, Brno
  - Research Site, Hradec Králové
  - Research Site, Prague
- France (7):
  - Research Site, Créteil
  - Research Site, Le Chesnay
  - Research Site, Nantes
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Pierre-Bénite
  - Research Site, Toulouse
- Germany (13):
  - Research Site, Berlin
  - Research Site, Cologne
  - Research Site, Essen
  - Research Site, Frankfurt am Main
  - Research Site, Freiburg im Breisgau
  - Research Site, Heidelberg
  - Research Site, Kiel
  - Research Site, Leipzig
  - Research Site, München
  - Research Site, Münster
  - Research Site, Tübingen
  - Research Site, Ulm
  - Research Site, Würzburg
- Greece (4):
  - Research Site, Athens
  - Research Site, Ioannina
  - Research Site, Pátrai
  - Research Site, Thessaloniki
- Research Site, Dublin, Ireland
- Israel (5):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Petah Tikva
  - Research Site, Tel Aviv
  - Research Site, Tel Litwinsky
- Italy (11):
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Bologna
  - Research Site, Florence
  - Research Site, Napoli
  - Research Site, Novara
  - Research Site, Palermo
  - Research Site, Roma
  - Research Site, Torino
  - Research Site, Venezia
  - Research Site, Verona
- Mexico (2):
  - Research Site, Mexico City, Mexico City
  - Research Site, Monterrey, Nuevo León
- Poland (3):
  - Research Site, Lublin
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Russia (4):
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Petrozavodsk
  - Research Site, Saratov
- South Korea (2):
  - Research Site, Busan
  - Research Site, Seoul
- Spain (5):
  - Research Site, Salamanca, Castille and León
  - Research Site, Badalona, Catalonia
  - Research Site, Oviedo, Principality of Asturias
  - Research Site, Valencia, Valencia
  - Research Site, Madrid
- Taiwan (4):
  - Research Site, Changhua
  - Research Site, Taichung
  - Research Site, Tainan
  - Research Site, Taipei
- Turkey (Türkiye) (4):
  - Research Site, Adana
  - Research Site, Ankara
  - Research Site, Istanbul
  - Research Site, Izmir
- United Kingdom (6):
  - Research Site, Bristol
  - Research Site, London
  - Research Site, Oxford
  - Research Site, Sheffield
  - Research Site, Southampton
  - Research Site, Sutton

REFERENCES:
- [Background] Delea TE, Amdahl J, Boyko D, Hagiwara M, Zimmerman ZF, Franklin JL, Cong Z, Hechmati G, Stein A. Cost-effectiveness of blinatumomab versus salvage chemotherapy in relapsed or refractory Philadelphia-chromosome-negative B-precursor acute lymphoblastic leukemia from a US payer perspective. J Med Econ. 2017 Sep;20(9):911-922. doi: 10.1080/13696998.2017.1344127. Epub 2017 Jul 11. PMID 28631497
- [Background] Kantarjian H, Stein A, Gokbuget N, Fielding AK, Schuh AC, Ribera JM, Wei A, Dombret H, Foa R, Bassan R, Arslan O, Sanz MA, Bergeron J, Demirkan F, Lech-Maranda E, Rambaldi A, Thomas X, Horst HA, Bruggemann M, Klapper W, Wood BL, Fleishman A, Nagorsen D, Holland C, Zimmerman Z, Topp MS. Blinatumomab versus Chemotherapy for Advanced Acute Lymphoblastic Leukemia. N Engl J Med. 2017 Mar 2;376(9):836-847. doi: 10.1056/NEJMoa1609783. PMID 28249141
- [Background] Dombret H, Topp MS, Schuh AC, Wei AH, Durrant S, Bacon CL, Tran Q, Zimmerman Z, Kantarjian H. Blinatumomab versus chemotherapy in first salvage or in later salvage for B-cell precursor acute lymphoblastic leukemia. Leuk Lymphoma. 2019 Sep;60(9):2214-2222. doi: 10.1080/10428194.2019.1576872. Epub 2019 Apr 5. PMID 30947585
- [Background] Kuchimanchi M, Zhu M, Clements JD, Doshi S. Exposure-response analysis of blinatumomab in patients with relapsed/refractory acute lymphoblastic leukaemia and comparison with standard of care chemotherapy. Br J Clin Pharmacol. 2019 Apr;85(4):807-817. doi: 10.1111/bcp.13864. Epub 2019 Feb 18. PMID 30645768
- [Background] Stein AS, Larson RA, Schuh AC, Stevenson W, Lech-Maranda E, Tran Q, Zimmerman Z, Kormany W, Topp MS. Exposure-adjusted adverse events comparing blinatumomab with chemotherapy in advanced acute lymphoblastic leukemia. Blood Adv. 2018 Jul 10;2(13):1522-1531. doi: 10.1182/bloodadvances.2018019034. PMID 29954814
- [Background] Topp MS, Zimmerman Z, Cannell P, Dombret H, Maertens J, Stein A, Franklin J, Tran Q, Cong Z, Schuh AC. Health-related quality of life in adults with relapsed/refractory acute lymphoblastic leukemia treated with blinatumomab. Blood. 2018 Jun 28;131(26):2906-2914. doi: 10.1182/blood-2017-09-804658. Epub 2018 May 8. PMID 29739753
- [Background] Kantarjian HM, Zugmaier G, Bruggemann M, Wood BL, Horst HA, Zeng Y, Martinelli G. Impact of Blinatumomab Treatment on Bone Marrow Function in Patients with Relapsed/Refractory B-Cell Precursor Acute Lymphoblastic Leukemia. Cancers (Basel). 2021 Nov 9;13(22):5607. doi: 10.3390/cancers13225607. PMID 34830762
- [Background] Horst HA, Zugmaier G, Martinelli G, Mergen N, Velasco K, Zaman F, Kantarjian H. CD19-negative relapse in adult patients with relapsed/refractory B-cell precursor acute lymphoblastic leukemia following treatment with blinatumomab-a post hoc analysis. Am J Hematol. 2023 Aug;98(8):E222-E225. doi: 10.1002/ajh.26988. Epub 2023 Jun 22. No abstract available. PMID 37345570
- [Derived] Shi Z, Zhu Y, Zhang J, Chen B. Monoclonal antibodies: new chance in the management of B-cell acute lymphoblastic leukemia. Hematology. 2022 Dec;27(1):642-652. doi: 10.1080/16078454.2022.2074704. PMID 35622074
- [Derived] Jabbour E, Patel K, Jain N, Duose D, Luthra R, Short NJ, Zugmaier G, San Lucas A, Velasco K, Tran Q, Zaman F, Konopleva M, Kantarjian H. Impact of Philadelphia chromosome-like alterations on efficacy and safety of blinatumomab in adults with relapsed/refractory acute lymphoblastic leukemia: A post hoc analysis from the phase 3 TOWER study. Am J Hematol. 2021 Oct 1;96(10):E379-E383. doi: 10.1002/ajh.26281. Epub 2021 Jul 7. No abstract available. PMID 34161631
- [Derived] Wei AH, Ribera JM, Larson RA, Ritchie D, Ghobadi A, Chen Y, Anderson A, Dos Santos CE, Franklin J, Kantarjian H. Biomarkers associated with blinatumomab outcomes in acute lymphoblastic leukemia. Leukemia. 2021 Aug;35(8):2220-2231. doi: 10.1038/s41375-020-01089-x. Epub 2021 Feb 4. PMID 33542479
- [Derived] Rambaldi A, Huguet F, Zak P, Cannell P, Tran Q, Franklin J, Topp MS. Blinatumomab consolidation and maintenance therapy in adults with relapsed/refractory B-precursor acute lymphoblastic leukemia. Blood Adv. 2020 Apr 14;4(7):1518-1525. doi: 10.1182/bloodadvances.2019000874. PMID 32289160
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 101 centers in 21 countries in Asia, Australia, Europe, and Latin and North America.
  The first participant was enrolled on 03 January 2014 and treated on 06 January 2014. The last participant enrolled on 25 September 2015 and the data cutoff date for this report was 04 January 2016.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to either blinatumomab or standard of care (SOC) chemotherapy regimens. Randomization was stratified by age (< 35 years vs ≥ 35 years), prior salvage therapy (yes vs no), and prior allogeneic hematopoietic stem cell transplantation (HSCT) (yes vs no) as assessed at the time of consent.
Period: Overall Study
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Started | 134 | 271
Received Treatment | 109 | 267
Completed | 33 (Indicates participants continuing study at time of data cut-off) | 93 (Indicates participants continuing study at time of data cut-off; 22 were receiving treatment)
Not Completed | 101 | 178
Not completed — Withdrawal by Subject | 15 | 14
Not completed — Sponsor Decision | 1 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Death | 85 | 160

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care Chemotherapy | Blinatumomab | Total
Number analyzed (Participants) | 134 | 271 | 405
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.1 (17.3) | 40.8 (17.1) | 40.9 (17.2)
Age, Customized [Number; unit: participants]
  < 35 years | 60 | 124 | 184
  35 to 54 years | 33 | 80 | 113
  55 to 64 years | 26 | 34 | 60
  ≥ 65 years | 15 | 33 | 48
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 109 | 166
  Male | 77 | 162 | 239
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 26 | 37
  Not Hispanic or Latino | 122 | 243 | 365
  Unknown or Not Reported | 1 | 2 | 3
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 4 | 5
  Asian | 9 | 19 | 28
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 3 | 5 | 8
  White | 112 | 228 | 340
  Multiple | 0 | 2 | 2
  Other | 8 | 12 | 20
Age Stratification at Randomization [Number; unit: participants]
  < 35 years | 60 | 123 | 183
  ≥ 35 years | 74 | 148 | 222
Prior Salvage Therapy Stratification at Randomization [Number; unit: participants]
  Yes | 80 | 164 | 244
  No | 54 | 107 | 161
Prior Allogeneic Hematopoietic Stem Cell Transplant (HCST) [Number; unit: participants]
  Yes | 46 | 94 | 140
  No | 88 | 177 | 265
Standard of Care Chemotherapy Regimen Received [Number; unit: participants] — FLAG = fludarabine, cytarabine arabinoside, and granulocyte colony-stimulating factor (filgrastim); HiDAC = high-dose cytarabine arabinoside
  participants
    FLAG ± anthracycline | 56 | 0 | 56
    High-dose methotrexate | 30 | 0 | 30
    Clofarabine | 26 | 0 | 26
    HIDAC | 22 | 0 | 22

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival
Description: Overall survival (OS) was calculated from time of randomization until death due to any cause. Participants still alive were censored at the date they were last known to be alive.
Time Frame: From randomization until the data cut-off date of 04 January 2016; median observation time was 11.8 months in the SOC group and 11.7 months in the blinatumomab group.
Population: All randomized participants
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
months | 4.0 [2.9 to 5.3] | 7.7 [5.6 to 9.6]
Statistical Analysis 1: Comparison: Standard of Care Chemotherapy vs Blinatumomab; Test type: Superiority or Other; p = 0.012, Stratified Log Rank; Stratified by age (< 35 years; ≥ 35 years), prior salvage therapy (yes vs. no), and prior allogeneic HSCT (yes vs. no); Hazard Ratio (HR) = 0.71, 95% CI 2-sided [0.55 to 0.93] — Hazard ratio obtained from the Cox Proportional Hazard Model. A hazard ratio < 1.0 indicated a lower average event rate and longer survival time for blinatumomab relative to SOC chemotherapy

2. Secondary Outcome: Percentage of Participants With Complete Remission Within 12 Weeks of Treatment Initiation
Description: Participants were evaluated for efficacy at the end of each treatment cycle via a central bone marrow aspiration and local peripheral blood counts.
  Complete Remission (CR) was defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts: platelets > 100,000/μl, and absolute neutrophil count (ANC) > 1,000/μl. CR must have occurred within 12 weeks of the first dose of therapy.
Time Frame: 12 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
percentage of participants | 15.7 [10.0 to 23.0] | 33.6 [28.0 to 39.5]
Statistical Analysis 1: Comparison: Standard of Care Chemotherapy vs Blinatumomab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; Adjusted for the stratification factors: age (< 35 vs. ≥ 35), prior salvage therapy (yes vs. no), and prior allogeneic HSCT (yes vs. no); Treatment difference = 17.9, 95% CI 2-sided [9.6 to 26.2]

3. Secondary Outcome: Percentage of Participants With Complete Remission/Complete Remission With Partial Hematological Recovery/Complete Remission With Incomplete Hematological Recovery (CR/CRh*/CRi) Within 12 Weeks of Treatment Initiation
Description: Participants were evaluated for efficacy at the end of each treatment cycle via a central bone marrow aspiration and local peripheral blood counts.
  Complete remission was defined as having ≤ 5% blasts in the bone marrow, no evidence of disease, and full recovery of peripheral blood counts: platelets > 100,000/μl, and ANC > 1,000/μl.
  Complete Remission with partial hematological recovery (CRh*) was defined as ≤ 5% blasts in the bone marrow, no evidence of disease and partial recovery of peripheral blood counts: platelets > 50,000/μl, and ANC > 500/μl.
  Complete remission with incomplete hematological recovery (CRi) was defined as ≤ 5% blasts in the bone marrow, no evidence of disease and incomplete recovery of peripheral blood counts: platelets > 100,000/μl or ANC > 1000 (but not both).
Time Frame: 12 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
percentage of participants | 24.6 [17.6 to 32.8] | 43.9 [37.9 to 50.0]
Statistical Analysis 1: Comparison: Standard of Care Chemotherapy vs Blinatumomab; Test type: Superiority or Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]; Treatment difference = 19.3, 95% CI 2-sided [9.9 to 28.7]

4. Secondary Outcome: Event Free Survival (EFS)
Description: Event free survival was defined as the time from randomization until a documented relapse after achieving CR/CRh*/CRi or death, whichever occurred first. Participants who failed to achieve a CR/CRh*/CRi within 12 weeks of treatment initiation were considered as non-responders and assigned an EFS duration of 1 day. Participants still alive and relapse-free were censored on their last disease assessment date.
  A relapse event was any one of the following:
  * Hematological relapse: proportion of blasts in bone marrow >5% or blasts in peripheral blood after documented CR or CRh* or CRi
  * Progressive disease: An increase from baseline of at least 25% of bone marrow blasts or an absolute increase of at least 5,000 cells/μL in the number of circulating leukemia cells
  * Extramedullary relapse: extramedullary lesion that is new or increased by 50% from nadir as assessed by Cheson criteria.
  The Kaplan-Meier estimate of EFS at 6 months is reported.
Time Frame: 6 months
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
percentage of participants | 12.5 [7.2 to 19.2] | 30.7 [25.0 to 36.5]
Statistical Analysis 1: Comparison: Standard of Care Chemotherapy vs Blinatumomab; Test type: Superiority or Other; Hazard Ratio (HR) = 0.55, 95% CI 2-sided [0.43 to 0.71] — The hazard ratio estimates were obtained from the Cox Proportional Hazard Model. A hazard ratio < 1.0 indicates a lower average event rate and a longer survival for Blinatumomab relative to SOC Chemotherapy

5. Secondary Outcome: Duration of Complete Remission
Description: Duration of complete remission, calculated only for participants who achieved a CR, was calculated from the date a CR was first achieved until the earliest date of a disease assessment indicating a relapse event or death, whichever occurred first. Participants who did not have a relapse event were censored on their last disease assessment date.
Time Frame: Up to the data cut-off date of 04 January 2016; median observation time was 10.8 months in the SOC group and 7.0 months in the blinatumomab group.
Population: Randomized participants with a best response of complete remission within 12 weeks of treatment initiation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 21 | 91
months | 7.8 [2.2 to 19.0] | 8.3 [5.7 to 10.7]

6. Secondary Outcome: Duration of Complete Remission/Complete Remission With Partial Hematological Recovery/Complete Remission With Incomplete Hematological Recovery (CR/CRh*/CRi)
Description: Duration of CR/CRh*/CRi, calculated only for participants who achieved a CR/CRh*/CRi, was calculated from the date a CR/CRh*/CRi was first achieved until the earliest date of a disease assessment indicating a relapse event or death, whichever occurred first. Participants who did not have a relapse event were censored on their last disease assessment date.
Time Frame: Up to the data cut-off date of 04 January 2016; median observation time was 10.8 months in the SOC group and 7.2 months in the blinatumomab group.
Population: Randomized participants with a best response of CR/CRh*/CRi within 12 weeks of treatment initiation.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 33 | 119
months | 4.6 [1.8 to 19.0] | 7.3 [5.8 to 9.9]

7. Secondary Outcome: Percentage of Participants With Minimal Residual Disease (MRD) Within 12 Weeks of Treatment Initiation
Description: Bone marrow samples were evaluated for MRD remission by a central laboratory. MRD remission was defined as the occurrence of an MRD level below 10^-4 measured by quantitative reverse transcription polymerase chain reaction (PCR) or flow cytometry.
Time Frame: 12 weeks
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
percentage of participants | 14.2 [8.8 to 21.3] | 29.9 [24.5 to 35.7]

8. Secondary Outcome: Percentage of Participants Who Received an Allogeneic Hematopoietic Stem Cell Transplant (HSCT)
Time Frame: Up to the data cut-off date of 04 January 2016; maximum time on study was 23 months.
Population: All randomized participants
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 134 | 271
percentage of participants | 23.9 [16.9 to 32.0] | 24.0 [19.0 to 29.5]

9. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events (AEs) were graded for severity according to the CTCAE version 4.0, where Grade 1: Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  Grade 2: Moderate; minimal, local or noninvasive intervention indicated; limiting age-appropriate instrumental activities of daily living.
  Grade 3: Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self care activities of daily living.
  Grade 4: Life-threatening consequences; urgent intervention indicated. Grade 5: Death related to AE. Treatment-related adverse events (TRAEs) were those assessed by the investigator as possibly related to blinatumomab based on response to the question: Is there a reasonable possibility that the event may have been caused by blinatumomab or other protocol-specified therapies/procedures?
Time Frame: From first dose of protocol-specified therapy until 30 days after the last dose, up to the data cut-off date of 04 January 2016; median duration of treatment was 5 days in the SOC group and 70 days in the blinatumomab group.
Population: All participants who received protocol-specified therapy analyzed according to the treatment they received.
Measure: Number; unit: participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 109 | 267
participants
  Any adverse event | 108 | 263
  AE grade ≥ 2 | 106 | 256
  AE grade ≥ 3 | 100 | 231
  AE grade ≥ 4 | 67 | 133
  Serious adverse events | 49 | 165
  AEs leading to interruption of study drug | 6 | 86
  AEs leading to discontinuation of study drug | 9 | 33
  Life-threatening adverse events | 26 | 55
  Fatal adverse events | 19 | 51
  Treatment-related adverse events | 92 | 214
  Treatment-related AE grade ≥ 2 | 89 | 195
  Treatment-related AE grade ≥ 3 | 78 | 143
  Treatment-related AE grade ≥ 4 | 51 | 57
  Serious treatment-related adverse events | 34 | 74
  TRAEs leading to interruption of study drug | 6 | 58
  TRAEs leading to discontinuation of study drug | 8 | 19
  Treatment-related life-threatening adverse events | 17 | 21
  Treatment-related fatal adverse events | 8 | 8

10. Secondary Outcome: 100-Day Mortality After Allogeneic Hematopoietic Stem Cell Transplant
Description: The analysis of 100-day mortality after allogeneic HSCT was assessed for participants who achieved a best response of CR/CRh*CTi within 12 weeks of treatment initiation, who received an allogeneic HSCT and did not receive any additional anticancer treatment before the transplant. 100-day mortality after allogeneic HSCT was calculated relative to the date of allogeneic HSCT.
  The 100-day mortality rate after allogeneic HSCT was defined as the percentage of participants having died up to 100 days after allogeneic HSCT estimated using the estimated time to death in percent calculated by Kaplan-Meier methods. Participants alive were censored on the last documented visit date or the date of the last phone contact when the patient was last known to have been alive.
Time Frame: 100 days, from the date of allogeneic HSCT until the data cut-off date of 04 January 2016
Population: Randomized participants with a best response of CR/CRh*/CRi within 12 weeks of treatment initiation and who received an allogeneic HSC without anti-cancer therapy prior to allogeneic HSCT.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 12 | 38
percentage of participants | 0.0 [NA to NA] — Could not be estimated due to the low number of events | 12.4 [4.8 to 29.9]

11. Secondary Outcome: Number of Participants With Anti-blinatumomab Antibodies
Description: Anti-blinatumomab binding antibodies were evaluated using a validated electrochemiluminescence (ECL)-based assay (binding assay). Samples positive for binding were analyzed using a cell-based bioassay to determine if the detected antibodies had neutralizing properties (neutralizing assay).
Time Frame: Samples were collected on day 29 at the end of cycle 2 and 30 days after the last dose of blinatumomab (median duration of treatment was 70 days).
Population: Participants who received blinatumomab with available post-baseline antibody data.
Measure: Number; unit: participants
Arm/Group | Blinatumomab
Number analyzed (Participants) | 171
participants
  Binding antibody positive | 5
  Neutralizing antibody positive | 3

12. Secondary Outcome: Time to a 10-point Decrease From Baseline in Global Health Status and Quality of Life or Death
Description: The European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) is a 30-item questionnaire that assesses the health related quality of life of cancer patients. The EORTC QLQ-C30 consists of a global health status/quality of life (QoL) scale, 5 functional scales, 3 symptom scales, and 6 single items.
  The global health/QoL scale consists of 2 questions that ask participants to rate their overall health and overall quality of life durig the past week on a scale from 1 (very poor) to 7 (excellent). The scale score was derived as the sum of each score and transformed to a scale from 0 to 100 where higher scores represent a high QoL.
  Time to a ≥10-point decrease from baseline GHS/QoL or death, whichever came first, was calculated from baseline. Participants still alive and without a 10-point decrease in GHS/QoL EORTC QLQ-C30 were censored on their last EORTC QLQ-C30 assessment date.
Time Frame: From randomization until the data cut-off date of 04 January 2016; EORTC QLQ-C30 was assessed on day 1, 8, 15, and 29 during cycle 1; days 1, 15, and 29 in cycle 2 and each consolidation cycle, and 30-days following the last dose of drug treatment.
Population: EORTC QLQ-C30 analysis set included all randomized participants with a non-missing baseline and at least 1 non-missing postbaseline result of any EORTC QLQ-C30 scales/item.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Number analyzed (Participants) | 95 | 247
months | 1.0 [0.5 to 1.5] | 1.7 [1.1 to 3.6]

ADVERSE EVENTS:
Time Frame: From first dose of protocol-specified therapy until 30 days after the last dose, up to the data cut-off date of 04 January 2016; median duration of treatment was 5 days in the SOC group and 70 days in the blinatumomab group.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | Standard of Care Chemotherapy | Blinatumomab
Serious Adverse Events (participants affected / at risk) | 49/109 | 165/267
Other Adverse Events (participants affected / at risk) | 105/109 | 250/267
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Chemotherapy (N=109) | Blinatumomab (N=267)
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 12 | 23
Histiocytosis haematophagic (Blood and lymphatic system disorders) | 0 | 3
Leukocytosis (Blood and lymphatic system disorders) | 0 | 3
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Aplasia (Congenital, familial and genetic disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Stomatitis (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Asthenia (General disorders) | 0 | 2
Chest pain (General disorders) | 0 | 1
Death (General disorders) | 0 | 1
Discomfort (General disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 2
Hyperthermia (General disorders) | 0 | 1
Medical device complication (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 4
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 16
Systemic inflammatory response syndrome (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 0 | 1
Acute graft versus host disease in skin (Immune system disorders) | 0 | 1
Anaphylactic shock (Immune system disorders) | 0 | 1
Cytokine release syndrome (Immune system disorders) | 0 | 7
Graft versus host disease (Immune system disorders) | 0 | 1
Graft versus host disease in liver (Immune system disorders) | 0 | 1
Abscess fungal (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 3 | 2
Bacterial infection (Infections and infestations) | 0 | 2
Bacterial sepsis (Infections and infestations) | 2 | 6
Brain abscess (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 4
Catheter site infection (Infections and infestations) | 0 | 2
Cellulitis (Infections and infestations) | 0 | 1
Central nervous system abscess (Infections and infestations) | 1 | 0
Citrobacter infection (Infections and infestations) | 0 | 1
Citrobacter sepsis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 6
Device related sepsis (Infections and infestations) | 2 | 1
Encephalitis enteroviral (Infections and infestations) | 0 | 1
Enterococcal bacteraemia (Infections and infestations) | 1 | 0
Enterococcal infection (Infections and infestations) | 1 | 0
Escherichia infection (Infections and infestations) | 0 | 2
Fungaemia (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 1 | 0
Fungal sepsis (Infections and infestations) | 0 | 2
Fusarium infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 2
Hepatosplenic candidiasis (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 0 | 1
Infection in an immunocompromised host (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lower respiratory tract infection fungal (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Meningitis bacterial (Infections and infestations) | 0 | 1
Mucormycosis (Infections and infestations) | 0 | 1
Muscle abscess (Infections and infestations) | 0 | 1
Neutropenic sepsis (Infections and infestations) | 1 | 3
Osteomyelitis (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 10
Pneumonia bacterial (Infections and infestations) | 0 | 1
Pneumonia fungal (Infections and infestations) | 2 | 1
Pneumonia pseudomonal (Infections and infestations) | 0 | 1
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 | 1
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 1
Pseudomonal sepsis (Infections and infestations) | 1 | 3
Pseudomonas infection (Infections and infestations) | 1 | 3
Pulmonary mycosis (Infections and infestations) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 7 | 13
Sepsis syndrome (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 3 | 8
Sinusitis (Infections and infestations) | 0 | 1
Skin infection (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal infection (Infections and infestations) | 1 | 2
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Streptococcal sepsis (Infections and infestations) | 1 | 0
Systemic candida (Infections and infestations) | 1 | 0
Tooth infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 3
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
Medication error (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 0 | 8
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 2
Blood lactate dehydrogenase increased (Investigations) | 0 | 1
CSF cell count abnormal (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
White blood cell count decreased (Investigations) | 0 | 1
White blood cell count increased (Investigations) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 2
Lactic acidosis (Metabolism and nutrition disorders) | 1 | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Osteitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemic infiltration extramedullary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Leukaemic infiltration pulmonary (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Aphasia (Nervous system disorders) | 0 | 3
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cognitive disorder (Nervous system disorders) | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 4
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 2 | 1
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Hemianopia (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hemiplegia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1
Intention tremor (Nervous system disorders) | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Neurological symptom (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 0 | 1
Status epilepticus (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 3
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Stridor (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1
Catheter placement (Surgical and medical procedures) | 0 | 1
Aortic occlusion (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 2 | 0
Peripheral artery thrombosis (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Standard of Care Chemotherapy (N=109) | Blinatumomab (N=267)
Anaemia (Blood and lymphatic system disorders) | 46 | 69
Febrile neutropenia (Blood and lymphatic system disorders) | 36 | 48
Neutropenia (Blood and lymphatic system disorders) | 31 | 51
Thrombocytopenia (Blood and lymphatic system disorders) | 32 | 47
Sinus tachycardia (Cardiac disorders) | 6 | 15
Tachycardia (Cardiac disorders) | 10 | 18
Abdominal pain (Gastrointestinal disorders) | 19 | 15
Constipation (Gastrointestinal disorders) | 28 | 34
Diarrhoea (Gastrointestinal disorders) | 38 | 58
Dyspepsia (Gastrointestinal disorders) | 7 | 10
Haemorrhoids (Gastrointestinal disorders) | 6 | 7
Nausea (Gastrointestinal disorders) | 46 | 51
Proctalgia (Gastrointestinal disorders) | 7 | 2
Stomatitis (Gastrointestinal disorders) | 14 | 17
Vomiting (Gastrointestinal disorders) | 26 | 31
Asthenia (General disorders) | 11 | 19
Chest pain (General disorders) | 6 | 6
Chills (General disorders) | 12 | 19
Fatigue (General disorders) | 14 | 34
Mucosal inflammation (General disorders) | 14 | 9
Oedema peripheral (General disorders) | 16 | 38
Pain (General disorders) | 6 | 16
Pyrexia (General disorders) | 48 | 153
Cytokine release syndrome (Immune system disorders) | 0 | 35
Hypogammaglobulinaemia (Immune system disorders) | 1 | 16
Bacteraemia (Infections and infestations) | 6 | 3
Oral herpes (Infections and infestations) | 9 | 15
Pneumonia (Infections and infestations) | 14 | 7
Sinusitis (Infections and infestations) | 6 | 5
Upper respiratory tract infection (Infections and infestations) | 1 | 19
Alanine aminotransferase increased (Investigations) | 11 | 24
Aspartate aminotransferase increased (Investigations) | 10 | 15
Blood bilirubin increased (Investigations) | 9 | 10
Neutrophil count decreased (Investigations) | 11 | 10
Platelet count decreased (Investigations) | 13 | 17
White blood cell count decreased (Investigations) | 6 | 13
Decreased appetite (Metabolism and nutrition disorders) | 15 | 18
Hyperglycaemia (Metabolism and nutrition disorders) | 9 | 20
Hypoalbuminaemia (Metabolism and nutrition disorders) | 11 | 13
Hypocalcaemia (Metabolism and nutrition disorders) | 9 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 30 | 45
Hypomagnesaemia (Metabolism and nutrition disorders) | 18 | 28
Hypophosphataemia (Metabolism and nutrition disorders) | 6 | 11
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 16
Back pain (Musculoskeletal and connective tissue disorders) | 10 | 33
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 29
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 19
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 25
Dizziness (Nervous system disorders) | 8 | 18
Headache (Nervous system disorders) | 32 | 77
Tremor (Nervous system disorders) | 0 | 26
Anxiety (Psychiatric disorders) | 6 | 13
Insomnia (Psychiatric disorders) | 10 | 28
Acute kidney injury (Renal and urinary disorders) | 6 | 8
Cough (Respiratory, thoracic and mediastinal disorders) | 6 | 39
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 15
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 9 | 16
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 7 | 13
Petechiae (Skin and subcutaneous tissue disorders) | 6 | 7
Rash (Skin and subcutaneous tissue disorders) | 13 | 19
Hypertension (Vascular disorders) | 9 | 17
Hypotension (Vascular disorders) | 11 | 32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.